CLINICAL TRIAL: NCT02424760
Title: A Prospective Cohort Study to Document the Clinical Outcomes in Shoulder Hemi-arthroplasty Using a PyC Spherical Interpositional Implant
Brief Title: Clinical Outcomes in Shoulder Hemi-arthroplasty Using a PyC Spherical Interpositional Implant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 0907-T-INSPYRE-RM
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2018-04

CONDITIONS: Localized, Primary Osteoarthritis; Post-traumatic Arthrosis of Other Joints, Shoulder Region; Avascular Necrosis of the Head of Humerus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Shoulder hemi-arthroplasty
  Other Names: Inspyre

SUMMARY:
The INSPYRE implant is a new range of shoulder hemi-arthroplasty device. It consists of a Pyrocarbon spherical interpositional implant and is indicated in primary surgery to relieve severe pain or significant disability caused by degenerative pathologies. The rotator cuff must be functional.

The aim of this study is to prospectively collect data from consecutive series to implement a Post Marketing Surveillance plan.

DETAILED DESCRIPTION:
Degenerative shoulder pathologies associated with a functional rotator cuff are currently treated by hemi-arthroplasty or total prosthesis replacement. The choice of surgery process is mainly made according to the status of the glenoid.

Concerning hemi-arthroplasty, two types of humeral prosthesis are usually used: anatomical stems or resurfacing head implants. Both provide good results. Nevertheless with these prostheses, patient can present with post-operative pains due to glenoid erosion, linked to the metallic compounds used in such a prostheses. To face this issue, it was decided to modify the metallic compounds, and in order to mimic the tribological properties of the cartilage, Pyrocarbon (PyC) was found to be the best material.

First application of PyC in a medical device was for cardiac valves in 1969. Currently more than 2 million people live with PyC cardiac valves. Mechanical and physical properties of PyC are in favor of its use in orthopedic surgery; furthermore, its biocompatibility plays an important role in its good acceptability.

As very good results were observed when used in hand and wrist, interposition PyC implant was suggested for shoulder. Another advantage was that such interposition device allowed performing less invasive surgery, a particularly important criteria for young patients.

INSPYRE shoulder prosthesis was then designed as a shoulder interposition implant intended for partial replacement of the gleno-humeral joint. This implant is inserted between the glenoid cartilage and the humeral metaphyseal cavity. It is indicated in primary surgery to relieve severe pain or significant disability caused by degenerative pathologies, e.g., osteoarthritis, rheumatoid arthritis, post-traumatic arthritis, primary and secondary necrosis of the humeral head. The rotator cuff must be functional.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring a Humeral Head Replacement (HHR) with INSPYRE as per indication of the Instruction For Use:
* with degenerative indication such as primary Gleno Humeral (GH) osteoarthritis, post-traumatic arthritis, primary and secondary avascular osteonecrosis of the humeral head,
* presenting a functional rotator cuff,
* able to return for all scheduled and required study visit;
* having provided informed Consent about scientific study participation if applicable.

Exclusion Criteria:

* Acute proximal humeral fracture,
* Systemic or local infection,
* Rotator cuff tear,
* Instability of the humeral head,
* Axillary nerve palsy,
* Revision arthroplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is a continuous series of the first 67 patients having received an Inspyre implant in the 8 participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-03; Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Implants survival rates | up to 10 years follow-up
  Number of device or procedure related adverse events

SECONDARY OUTCOMES:
Change from baseline and previous visit in Constant Murley score | at 1, 2, 5 and 10 years follow-up
Change from baseline and previous visit in Range of Motion | at 3-6 months, 1, 2, 5 and 10 years follow-up
  Forward flexion, Internal rotation and external rotation will be assessed
Radiographic criteria timely evolution | at 3-6 months, 1, 2, 5 and 10 years follow-up
  Glenoid erosion, tuberosities thinning, lateralization index, subacromial space and implant subsidence will be assessed according to available R-ray, CT or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Gilles WALCH, MD, Principal Investigator — Centre Orthopédique Santy, Lyon, FR